CLINICAL TRIAL: NCT03611153
Title: Hemodynamic Effects of a Novel Myeloperoxidase Inhibitor With Exercise in Heart Failure With Preserved Ejection Fraction - A Randomized, Double-Blind, Placebo Controlled Proof of Principle Study
Brief Title: Myeloperoxidase (MPO) Inhibitor A_Zeneca for Heart Failure With Preserved Ejection Fraction (HFpEF)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Barry Borlaug, Principle Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17-002907; UL1TR000135 (NIH)
Record Dates: First submitted 2018-07-26; First posted 2018-08-02 (Actual); Results first posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: Heart Failure
Keywords: Heart Failure; Ejection Fraction; Preserved; Myeloperoxidase Inhibitor; Exercise
MeSH Terms: conditions — Heart Failure; Motor Activity

STUDY DESIGN:
Intervention Model Description: Single Administration of study drug
Who Masked: Participant, Investigator
Masking Description: Only research pharmacy staff will be aware of randomization scheme and all study personnel and subjects will remain blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AZD4831 Oral myeloperoxidase inhibitor (Experimental): Patient may take 30 mg of oral myeloperoxidase inhibitor following baseline right heart catheterization.
  Interventions: Drug: AZD4831 Oral Myeloperoxidase Inhibitor
- Placebo (Placebo Comparator): Patient may take 30 mg of placebo oral capsule following baseline right heart catheterization.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: AZD4831 Oral Myeloperoxidase Inhibitor — A single administration dose of 30 mg oral MPO inhibitor given orally following baseline, resting and exercise testing in patients during right heart catheterization.
  Other Names: Oral MPO inhibitor AZD4831
  Arms: AZD4831 Oral myeloperoxidase inhibitor
Drug: Placebo oral capsule — A single administration dose of 30 mg placebo given orally following baseline, resting and exercise testing in patients during right heart catheterization.
  Arms: Placebo

SUMMARY:
Researchers are studying the effect of a single dose of oral myeloperoxidase on heart failure versus placebo.

DETAILED DESCRIPTION:
Enroll subjects with a normal ejection fraction referred to the catheterization laboratory for evaluation of breathlessness or shortness of breath. Perform safety lab sampling, echocardiography, arterial tonometry for pulse wave analysis, and assessment of endothelial function prior to administration of study drug. During the catheterization researchers will perform blood draws, assess baseline exercise capacity at rest and during exercise. Researchers will also do an echocardiogram to take measurements of the heart. Subjects will be randomized to one of two groups, Oral Myeloperoxidase Inhibitor or placebo group. Study drug or placebo will be administered followed by a repeat of the baseline catheterization assessments. At the conclusion of the second exercise test the subject will be moved to a room and monitored overnight for safety. Repeat blood draws, echocardiogram, endothelial function test, and heart monitoring will be completed. The subject will be asked to follow up with the researchers between 9-14 days after the study drug dosage. The subjects history and blood work will be completed at that visit.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females of non-childbearing potential
2. Age ≥ 30 years
3. Symptoms of dyspnea (II-IV) at the time of screening
4. Ejection Fraction (EF) ≥ 50% as determined on imaging study within 12 months of enrollment
5. Catheterization documented elevated filling pressures at rest (PCWP ≥15) or with exercise (PCWP ≥25)

Exclusion Criteria:

1. Use of nitrates, phosphodiesterase 5 inhibitors or other NO-providing therapy in the past 24 hours of screening
2. Significant valvular disease (>moderate left-sided regurgitation, >mild stenosis)
3. Requirement of intravenous heparin at the start of case
4. Severe pulmonary parenchymal disease
5. Acute coronary syndrome or coronary disease requiring revascularization in the judgement of investigators
6. Resting systolic blood pressure < 100 mmHg
7. Constrictive pericarditis
8. Infiltrative, restrictive, or hypertrophic obstructive cardiomyopathies
9. Previous anaphylaxis to any drug
10. Pregnancy or breastfeeding mothers
11. High Output heart failure
12. Active thyroid disease
13. Treatment with a new chemical entity (defined as a compound which has not been approved for marketing) within the preceding 3 months
14. Patients with any prior allergy to propylthiouracil

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2022-02-11 (Actual); Study Completion 2022-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barry A Borlaug, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- AZD4831 Oral Myeloperoxidase Inhibitor: Patient may take 30 mg of oral myeloperoxidase inhibitor following baseline right heart catheterization.
  AZD4831 Oral Myeloperoxidase(MPO) Inhibitor: A single administration dose of 30 mg oral MPO inhibitor given orally following baseline, resting and exercise testing in patients during right heart catheterization.
Period: Overall Study
Arm/Group | AZD4831 Oral Myeloperoxidase Inhibitor | Placebo
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD4831 Oral Myeloperoxidase Inhibitor | Placebo | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (12) | 70 (6) | 70 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 10 | 9 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 15 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 15 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Change in Exercise Pulmonary Capillary Wedge Pressure (PCWP)
Description: Pulmonary capillary wedge pressure (PCWP) provides an indirect estimate of left atrial pressure (LAP). PCWP is the pressure measured by wedging a pulmonary catheter with an inflated balloon into a small pulmonary arterial branch. The exercise PCWP values are obtained at 20 Watt workload, measured in mmHg.
Time Frame: Baseline, approximately 30 minutes after study drug administration
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AZD4831 Oral Myeloperoxidase Inhibitor | Placebo
Number analyzed (Participants) | 15 | 15
mmHg | -1 (3) | -4 (5)
Statistical Analysis 1: Comparison: AZD4831 Oral Myeloperoxidase Inhibitor vs Placebo; Test type: Superiority; p = 0.040, ANCOVA

2. Primary Outcome: Exercise Pulmonary Capillary Wedge Pressure (PCWP)
Description: as for outcome 1
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AZD4831 Oral Myeloperoxidase Inhibitor | Placebo
Number analyzed (Participants) | 15 | 15
mmHg | 31 (6) | 32 (7)

3. Secondary Outcome: Change in Resting Pulmonary Capillary Wedge Pressure (PCWP)
Description: Pulmonary capillary wedge pressure (PCWP) provides an indirect estimate of left atrial pressure (LAP). PCWP is the pressure measured by wedging a pulmonary catheter with an inflated balloon into a small pulmonary arterial branch while in resting state, measured in mmHg.
Time Frame: Baseline, approximately 30 minutes after study drug administration
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AZD4831 Oral Myeloperoxidase Inhibitor | Placebo
Number analyzed (Participants) | 15 | 15
mmHg | -2 (3) | -2 (2)
Statistical Analysis 1: Comparison: AZD4831 Oral Myeloperoxidase Inhibitor vs Placebo; Test type: Superiority; p = 0.777, t-test, 2 sided

4. Secondary Outcome: Change in Exercise Central Pressures
Description: Exercise values after receiving study drug minus exercise values before study drug, obtained at 20 Watt workload, measured in mmHg.
Time Frame: Baseline, approximately 30 minutes after study drug administration
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AZD4831 Oral Myeloperoxidase Inhibitor | Placebo
Number analyzed (Participants) | 15 | 15
mmHg
  Right atrial pressure | 0 (3) | 0 (2)
  Pulmonary artery systolic pressure | -2 (5) | -4 (5)
  Mean pulmonary artery pressure | -1 (4) | -4 (5)
Statistical Analysis 1: Comparison: AZD4831 Oral Myeloperoxidase Inhibitor vs Placebo; Right atrial pressure; Test type: Superiority; p = 0.805, t-test, 2 sided
Statistical Analysis 2: Comparison: AZD4831 Oral Myeloperoxidase Inhibitor vs Placebo; pulmonary artery systolic pressure; Test type: Superiority; p = 0.148, t-test, 2 sided
Statistical Analysis 3: Comparison: AZD4831 Oral Myeloperoxidase Inhibitor vs Placebo; Mean pulmonary artery pressure; Test type: Superiority; p = 0.090, t-test, 2 sided

5. Secondary Outcome: Change in Resting Central Pressures
Description: Resting values after receiving study drug minus resting values before study drug, measured in mmHg.
Time Frame: Baseline, approximately 30 minutes after study drug administration
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AZD4831 Oral Myeloperoxidase Inhibitor | Placebo
Number analyzed (Participants) | 15 | 15
mmHg
  Right atrial pressure | 0 (2) | 0 (1)
  Pulmonary artery systolic pressure | -3 (5) | -3 (5)
  Mean pulmonary artery pressure | -1 (3) | -2 (3)
Statistical Analysis 1: Comparison: AZD4831 Oral Myeloperoxidase Inhibitor vs Placebo; Right atrial pressure; Test type: Superiority; p = 0.786, t-test, 2 sided
Statistical Analysis 2: Comparison: AZD4831 Oral Myeloperoxidase Inhibitor vs Placebo; Pulmonary artery systolic pressure; Test type: Superiority; p = 0.796, t-test, 2 sided
Statistical Analysis 3: Comparison: AZD4831 Oral Myeloperoxidase Inhibitor vs Placebo; Mean pulmonary artery pressure; Test type: Superiority; p = 0.703, t-test, 2 sided

6. Secondary Outcome: Change in Exercise Transmyocardial Lactate Ratio
Description: Obtained at 20 Watt workload, determined by the lactate extraction ratio, which is calculated as lactate arterial minus lactate coronary sinus (CS) divided by lactate arterial. Negative values are indicative of myocardial ischemia.
Time Frame: Baseline, approximately 30 minutes after drug administration
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | AZD4831 Oral Myeloperoxidase Inhibitor | Placebo
Number analyzed (Participants) | 15 | 15
ratio | 0.05 (0.17) | -0.01 (0.15)
Statistical Analysis 1: Comparison: AZD4831 Oral Myeloperoxidase Inhibitor vs Placebo; Test type: Superiority; p = 0.418, t-test, 2 sided

7. Secondary Outcome: Change in Resting Transmyocardial Lactate Ratio
Description: Obtained during resting state, determined by the lactate extraction ratio, which is calculated as lactate arterial minus lactate coronary sinus (CS) divided by lactate arterial. Negative values are indicative of myocardial ischemia.
Time Frame: Baseline, approximately 30 minutes after drug administration
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | AZD4831 Oral Myeloperoxidase Inhibitor | Placebo
Number analyzed (Participants) | 15 | 15
ratio | 0.16 (0.49) | 0.10 (0.23)
Statistical Analysis 1: Comparison: AZD4831 Oral Myeloperoxidase Inhibitor vs Placebo; Test type: Superiority; p = 0.669, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events were collected on each participant from the start of the invasive testing procedure and study drug administration, through the follow-up visit, which was approximately 9-14 days later; for a total of approximately 15 days.
Arm/Group | AZD4831 Oral Myeloperoxidase Inhibitor | Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 1/15
Other Adverse Events (participants affected / at risk) | 2/15 | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD4831 Oral Myeloperoxidase Inhibitor (N=15) | Placebo (N=15)
Hospitalization for Heart Failure (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD4831 Oral Myeloperoxidase Inhibitor (N=15) | Placebo (N=15)
Nausea (General disorders) | 1 (1) | 0 (0)
Vomiting (General disorders) | 1 (1) | 0 (0)
Diarrhea (General disorders) | 1 (1) | 0 (0)
Lower extremity deep vein thrombosis (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-11): https://cdn.clinicaltrials.gov/large-docs/53/NCT03611153/Prot_SAP_000.pdf